

MoveLab; Physical Activity and Exercise Research Faculty of Medical Sciences 4<sup>th</sup> Floor William Leech Building Newcastle University Newcastle upon Tyne NE2 4HH T: +44 (0)191 222 8264

The Newcastle upon Tyne Hospitals NHS
NHS Foundation Trust

Patient Identification number for this trial:

## **CONSENT FORM**

Title of Project: Physical Activity in Heart Failure

Name of researchers: Dr Djordje Jakovljevic, Dr Jane Skinner, Dr Guy MacGowan, Dr Kristian Bailey, Dr Sarah Moore, Dr Leah Avery, Dr Nicki O'Brien, Dr Christopher Eggett

| | | | Please | initial box |
|---|---|---|---|---|
| 1. | | ave read and understand the information sheet dated 4 <sup>th</sup> April D) for the above study and have had the opportunity to ask | | |
| 2. | understand that my participant is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | I agree to my GP being informed of my participation in the study. | | | |
| 4. | I understand that my results will be kept confidential. | | | |
| 5. | I understand that my data will be stored securely. | | | |
| 6. | I understand that relevant sections of my medical notes and data collected during the study,may be looked at by members of the research team or individuals from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 7. | I agree to take part in the above study. | | | |
| | I agree, that if asked I will take pumber of the research team and orpose of this research. | | | |
| —<br>Nan | ne of patient | Date | Signature | |
| Name of person taking consent (if different from researcher) | | Date | Signature | |
| Researcher | | <br>Date | <br>Signature | |

1 copy for patient; 1 copyt for researcher; 1 copy to be kept within medical records